CLINICAL TRIAL: NCT03739034
Title: Evaluation of a Lifestyle Medicine Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, David Drozek, Associate Professor, Ohio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-X-220
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Chronic Lifestyle Related Disease; Diabetes; Overweight and Obesity; Dyslipidemias; Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus; Overweight; Obesity; Dyslipidemias; Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients are being treated with established lifestyle medicine modalities, tailored to the individual patient need and situation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Medicine (Experimental): Patients presenting for lifestyle medicine treatment to prevent, arrest or reverse chronic lifestyle related diseases.
  Interventions: Behavioral: Lifestyle Medicine

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Treatment modalities consist of encouraging a plant based, whole food diet, physical activity, stress management, healthy sleep, control of unhealthy habits.

SUMMARY:
This project will evaluate the success of the PI's lifestyle medicine practice.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the effectiveness of the PI's lifestyle medicine practice over time.

Sub-objectives are:

1. Understand variables that affect success in application of lifestyle medicine to lead to improved patient outcomes.
2. Develop a model for practice evaluation that can be utilized for board certification of providers and practices that utilize lifestyle medicine.
3. Evaluate the reimbursement success of lifestyle medicine services as a factor of billing codes and insurance providers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are seen by the PI in his lifestyle medicine practice at Muntean Health Care.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Weight | 1 year
  change in weight
Systolic Blood Pressure | 1 year
  change in systolic blood pressure
Diastolic Blood Pressure | 1 year
  change in diastolic blood pressure
Glycosylated hemoglobin | 1 year
  change in glycosylated hemoglobin
Total cholesterol | 1 year
  change in total cholesterol
low density lipoprotein cholesterol | 1 year
  change in low density lipoprotein cholesterol
triglycerides | 1 year
  change in triglycerides
high density lipoprotein cholesterol | 1 year
  change in high density lipoprotein cholesterol

SECONDARY OUTCOMES:
steps | 1 year
  average number of steps per day
exercise | 1 year
  average minutes of exercise per day
fiber | 1 year
  average grams of fiber consumed on a daily basis
legumes | 1 year
  average quantity of legumes consumed on a daily basis
full plate | 1 year
  average percent of plate filled with foods high in fiber and water

CONTACTS AND LOCATIONS:
Overall Officials: David S Drozek, DO, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No